CLINICAL TRIAL: NCT07101224
Title: Data Registry in Chinese Hemophilia A and B Patients Related to the Use of Anti-hemophilic Coagulation Factor Replacement Therapy
Brief Title: Data Registry in Chinese Hemophilia A and B Patients
Status: Completed | Type: Observational
Sponsor: Institute of Hematology & Blood Diseases Hospital, China (Other)
Responsible Party: Sponsor
Other Study IDs: QT2016004
Record Dates: First submitted 2017-05-26; First posted 2025-08-03 (Actual); Last update posted 2025-08-03 (Actual); Status verified 2024-05

CONDITIONS: Hemophilia A; Hemophilia B
Keywords: anti-hemophilic coagulation factor replacement therapy
MeSH Terms: conditions — Hemophilia A; Hemophilia B

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 2 Years
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

GROUPS / COHORTS (2):
- Hemophilia A
- Hemophilia B

SUMMARY:
This is an open-label, prospective, multi-center, patient registry in Chinese Hemophilia A and B patients treated with anti-hemophilic coagulation factor replacement therapy.

ELIGIBILITY:
Inclusion Criteria：

Subjects must meet all of the following inclusion criteria to be eligible for enrollment into the study:

1. Hemophilia A and Hemophilia B patient diagnosed;
2. Taking anti-hemophilic coagulation factor replacement therapy during the 2 year registry period.

Exclusion Criteria:

1. Unwilling or unable to follow the terms of the protocol.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: Diagnosed Hemophilia A and Hemophilia B patient with anti-hemophilic coagulation factor replacement therapy will be selected.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2017-05-07 (Actual); Primary Completion 2019-06-30 (Actual); Study Completion 2019-06-30 (Actual)

PRIMARY OUTCOMES:
The incidence of MIEs and other SAEs | at the end of 2 year data registry
  The incidence of MIE(medically important events)s and other SAE(serious adverse event)s in the anti-hemophilic replacement treatment

SECONDARY OUTCOMES:
Treatment regimen | at the end of 2 year data registry
  Treatment regimen of anti-hemophilic replacement treatment

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital of Blood disease, Tianjin, Tianjin Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided